CLINICAL TRIAL: NCT03788239
Title: Wound Closure After Total Knee Replacement: Comparison Between Staples and Sutures.
Brief Title: Wound Closure After Total Knee Replacement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Indus Hospital and Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRD_IRB_2017_06_006
Record Dates: First submitted 2018-12-24; First posted 2018-12-27 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Wound of Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Right knee wound closure by staples and Left Knee wound closure by sutures
  Interventions: Other: Staples versus sutures
- Arm 2 (Experimental): Right knee wound closure by sutures and Left Knee wound closure by staples
  Interventions: Other: Staples versus sutures

INTERVENTIONS:
Other: Staples versus sutures — Prolene suture: non-absorbable, sterile surgical suture composed of an isotactic crystalline steroisomer of polypropylene, a synthetic linear polyolefin. After completion of the procedure, deep tissues will closed with subcuticular prolene suture. Compared to the absorbable sutures, prolene is known to cause less infection since it is a monofilament material.
  Staples: specialized staples used in surgery in place of sutures to close skin wounds. After completion of the procedure, deep tissues were closed with absorbable braided suture, then the skin will be closed by staples.

SUMMARY:
To compare the wound healing after total knee replacement wound closure with staples versus subcuticular prolene suture.

DETAILED DESCRIPTION:
.Informed consent will be taken from all the patients who meet the inclusion and exclusion criteria and then will be randomized into one of the two study arms (Arm 1: will undergo wound closure with staples and Arm 2 wound closure with subcuticular prolene suture).

before the start of surgery. The primary investigator will open the sealed envelopes provided by the Indus Hospital Research Center's Clinical Research Unit (CRU) that provides the study arm allocation. The envelopes will follow the SNOSE protocol i.e. they will be sequentially numbered, opaque sealed envelopes. Before opening the envelope, the primary investigator will write the patient's medical record number, date and will sign the envelope. The envelope will contain carbon paper which will transfer the data allocation paper inside.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary total knee replacements for osteoarthritis or post-traumatic arthritis (diagnosed on X-rays and history)
* Bilateral knee surgeries
* Patients giving informed consent

Exclusion Criteria:

* Patients having previous skin, neuromuscular or connective tissue disorder (confirmed by history)
* Patients taking steroids (confirmed by history)
* Body mass index > 30 (increases chances of wound dehiscence)
* Lack of consent
* Pregnant females (confirmed by history)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Wound healing | Surgery till 1 year post-op
  Wound healing will be assessed using Hollander Score
Complications | Surgery till 1 year post-op

CONTACTS AND LOCATIONS:
Locations (1):
- The Indus Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided